CLINICAL TRIAL: NCT01652716
Title: A Randomized, Open-Label, Long-Term, Parallel-Group, Comparator-Controlled, Multicenter Study to Compare the Glycemic Effects, Safety, and Tolerability of Exenatide Once Weekly Suspension to Exenatide Twice Daily in Subjects With Type 2 Diabetes Mellitus
Brief Title: Efficacy and Safety of Exenatide Once Weekly Suspension in Subjects With Type 2 Diabetes
Acronym: DURATION-NEO-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCB118; MB001-003 (Other: Bristol Myers Squibb)
Record Dates: First submitted 2012-07-26; First posted 2012-07-30 (Estimated); Results first posted 2015-09-16 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exenatide once weekly suspension (Experimental): Exenatide suspension 2 mg weekly subcutaneous injection
  Interventions: Drug: Exenatide once weekly suspension
- Exenatide twice daily (BID) (Active Comparator): Exenatide 5 mcg BID for 4 weeks followed by 10 mcg BID for 24 weeks
  Interventions: Drug: Exenatide twice daily

INTERVENTIONS:
Drug: Exenatide once weekly suspension — Exenatide suspension 2 mg weekly subcutaneous injection
  Arms: Exenatide once weekly suspension
Drug: Exenatide twice daily — 5 mcg twice daily for 4 weeks followed by 10 mcg twice daily for 24 weeks
  Other Names: Byetta
  Arms: Exenatide twice daily (BID)

SUMMARY:
To compare the effect on glycemic control (HbA1c) of exenatide suspension administered once weekly to that achieved by exenatide administered twice daily for 28 weeks in subjects with type 2 diabetes mellitus.

To examine the long-term (52 weeks of treatment) safety and effect on glucose control of exenatide suspension administered once weekly in subjects with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Diagnosed with type 2 diabetes mellitus
* HbA1c 7.1 to 11%, inclusive, at screening
* Fasting plasma glucose <280 mg/dL (15.5 mmol/L)
* Body mass index (BMI) <=45 kg/m2, inclusive, at screening
* Treated with diet and exercise or a stable regimen of metformin, sulfonylurea, pioglitazone or any 2 of these agents

Exclusion Criteria:

* History of pancreatitis or triglycerides >=500 mg/dL
* Medullary carcinoma or multiple endocrine neoplasia (MEN2) or a family history of either
* Active cardiovascular disease
* Presence of congestive heart failure
* Liver disease
* History of severe gastrointestinal diseases
* Repeated severe hypoglycemia within the last 6 months
* Any previous use of exenatide or other glucagon-like peptide-1 (GLP-1 ) analog
* Dipeptidyl peptidase-4 (DPP-4) inhibitor use in the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 377 (Actual)
Dates: Start 2013-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vice President Medical Research & Development, M.D., Study Director — Amylin Pharmaceuticals, LLC.
Locations (55):
- United States (55):
  - Research Site, Muscle Shoals, Alabama
  - Research Site, Mesa, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Escondido, California
  - Research Site, Garden Grove, California
  - Research Site, Lomita, California
  - Research Site, Los Angeles, California
  - Research Site, Santa Ana, California
  - Research Site, Spring Valley, California
  - Research Site, Walnut Creek, California
  - Research Site, Denver, Colorado
  - Research Site, Coral Gables, Florida
  - Research Site, DeLand, Florida
  - Research Site, Kissimmee, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Oviedo, Florida
  - Research Site, Palm Harbor, Florida
  - Research Site, Ponte Vedra, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Lexington, Kentucky
  - Research Site, Paducah, Kentucky
  - Research Site, Lake Charles, Louisiana
  - Research Site, Columbia, Maryland
  - Research Site, Elkridge, Maryland
  - Research Site, Hyattsville, Maryland
  - Research Site, New Bedford, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Troy, Michigan
  - Research Site, Edina, Minnesota
  - Research Site, Port Gibson, Mississippi
  - Research Site, St Louis, Missouri
  - Research Site, Butte, Montana
  - Research Site, Henderson, Nevada
  - Research Site, Endwell, New York
  - Research Site, New Windsor, New York
  - Research Site, Greensboro, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Portland, Oregon
  - Research Site, Harleysville, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Murray, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, Manassas, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Olympia, Washington
  - Research Site, Spokane, Washington

REFERENCES:
- [Derived] Wysham CH, Rosenstock J, Vetter ML, Wang H, Hardy E, Iqbal N. Further improvement in glycemic control after switching from exenatide two times per day to exenatide once-weekly autoinjected suspension in patients with type 2 diabetes: 52-week results from the DURATION-NEO-1 study. BMJ Open Diabetes Res Care. 2020 Oct;8(1):e000773. doi: 10.1136/bmjdrc-2019-000773. PMID 33037036
- [Derived] Wysham CH, Rosenstock J, Vetter ML, Dong F, Ohman P, Iqbal N. Efficacy and tolerability of the new autoinjected suspension of exenatide once weekly versus exenatide twice daily in patients with type 2 diabetes. Diabetes Obes Metab. 2018 Jan;20(1):165-172. doi: 10.1111/dom.13056. Epub 2017 Aug 22. PMID 28685973

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were randomized across two treatment groups (exenatide once weekly and exenatide twice daily) in a ratio of 3:2 with randomization stratified by diabetes management method at screening, screening haemoglobin A1c (HbA1c) stratum and renal function.
Groups:
- Experimental: Exenatide Once Weekly (QWS) Suspension: Exenatide suspension 2 mg weekly subcutaneous injection for 52 weeks (28 weeks plus an additional 24 weeks)
- Active Comparator: Exenatide Twice Daily (BID): Exenatide 5 mcg BID for 4 weeks followed by 10 mcg BID for 24 weeks followed by a switch to Exenatide QWS 2mg for at least 24 weeks
Period: Overall Study
Arm/Group | Experimental: Exenatide Once Weekly (QWS) Suspension | Active Comparator: Exenatide Twice Daily (BID)
Started | 229 | 148 (Two subjects in the exenatide BID group withdrew from the study before receiving study drug.)
Completed 28-week | 197 | 118
Completed | 173 (* completed study) | 102 (* completed study)
Not Completed | 56 | 46
Not completed — Loss of glucose control | 1 | 0
Not completed — Administrative | 0 | 2
Not completed — Investigator decision | 1 | 4
Not completed — Lost to Follow-up | 12 | 11
Not completed — Protocol Violation | 2 | 1
Not completed — Adverse Event | 7 | 10
Not completed — Withdrawal by Subject | 33 | 18

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-Treat: Subjects who were randomized and received at least one dose of study drug
Groups:
- Experimental: Exenatide QWS Suspension: Exenatide suspension 2 mg weekly subcutaneous injection 52 weeks (28 weeks plus an additional 24 weeks)
- Active Comparator: Exenatide BID: Exenatide 5 mcg BID for 4 weeks followed by 10 mcg BID for 24 weeks followed by a switch to Exenatide QWS 2mg for at least 24 weeks
- Total: Total of all reporting groups
Arm/Group | Experimental: Exenatide QWS Suspension | Active Comparator: Exenatide BID | Total
Number analyzed (Participants) | 229 | 146 | 375
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.6 (9.98) | 56.5 (9.04) | 56.0 (9.62)
Age, Customized [Number; unit: Participants]
  <65 years | 182 | 118 | 300
  >=65 years | 47 | 28 | 75
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 54 | 135
  Male | 148 | 92 | 240
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 54 | 34 | 88
  Not Hispanic or Latino | 174 | 112 | 286
  Unknown | 1 | 0 | 1
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 168 | 110 | 278
  Black or African American | 38 | 23 | 61
  Asian | 17 | 8 | 25
  Other | 3 | 2 | 5
  American Indian or Alaska Native | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
Weight [Mean (Standard Deviation); unit: lbs] | 214.52 (49.788) | 213.19 (40.834) | 214.00 (46.445)
Baseline HbA1c [Mean (Standard Deviation); unit: Percentage of total hemoglobin] | 8.47 (1.047) | 8.51 (1.004) | 8.48 (1.029)
HbA1c Stratum [Number; unit: Number of subjects]
  <9.0% | 159 | 97 | 256
  >=9.0% | 68 | 49 | 117
  Not Recorded | 2 | 0 | 2
Fasting plasma glucose [Mean (Standard Deviation); unit: mg/dL] | 180.92 (44.538) | 183.77 (46.904) | 182.03 (45.437)
Duration of diabetes [Mean (Standard Deviation); unit: Years] | 8.55 (6.249) | 8.47 (5.961) | 8.52 (6.132)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c (Glycosylated Hemoglobin) From Baseline to Week 28
Description: The primary objective of this study was to compare the effect on glycemic control (HbA1c) of exenatide suspension administered once weekly to that achieved by exenatide administered twice daily for 28 weeks in subjects with type 2 diabetes mellitus.
Time Frame: Baseline to Week 28
Population: Modified Intent-to-Treat: Subjects who were randomized and received at least one dose of study drug
Measure: Least Squares Mean (Standard Error); unit: Percentage of total hemoglobin
Arm/Group | Experimental: Exenatide QWS Suspension | Active Comparator: Exenatide BID
Number analyzed (Participants) | 229 | 146
Percentage of total hemoglobin | -1.39 (0.0930) | -1.02 (0.1147)
Statistical Analysis 1: Comparison: Experimental: Exenatide QWS Suspension vs Active Comparator: Exenatide BID; Test type: Superiority or Other; p = 0.0072, Mixed model for repeated measure (MMRM); Based on a repeated measures mixed model including fixed categorical effects of treatment; LS Mean Difference = -0.37, 95% CI 2-sided [-0.63 to -0.10], Standard Error of Mean 0.1349

2. Secondary Outcome: Percentage of Subjects Achieving HbA1c <7% at Week 28
Description: Percentage of subjects achieving HbA1c <7% at Week 28/Study Termination
Time Frame: Baseline to Week 28
Population: Modified Intent-to-Treat: Subjects who were randomized and received at least one dose of study drug.
Measure: Number; unit: Percentage of subjects
Arm/Group | Experimental: Exenatide QWS Suspension | Active Comparator: Exenatide BID
Number analyzed (Participants) | 229 | 146
Percentage of subjects
  Baseline Yes | 3.9 | 1.4
  Baseline No | 95.2 | 98.6
  Week 28 Yes | 49.3 | 43.2
  Week 28 No | 49.8 | 56.8
  Baseline missing | 0.9 | 0
Statistical Analysis 1: Comparison: Experimental: Exenatide QWS Suspension vs Active Comparator: Exenatide BID; Test type: Superiority or Other; p = 0.2247, Cochran-Mantel-Haenszel

3. Secondary Outcome: Change in Fasting Plasma Glucose Concentrations From Baseline to Week 28
Description: Change in fasting plasma glucose concentrations from baseline to Week 28/Study Termination
Time Frame: Baseline to Week 28
Population: Modified Intent-to-Treat: Subjects who were randomized and received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Experimental: Exenatide QWS Suspension | Active Comparator: Exenatide BID
Number analyzed (Participants) | 229 | 146
mg/dL | -32.7 (3.906) | -22.5 (4.917)
Statistical Analysis 1: Comparison: Experimental: Exenatide QWS Suspension vs Active Comparator: Exenatide BID; Test type: Superiority or Other; p = 0.1656, Cochran-Mantel-Haenszel — Adjusted; LS Mean Difference = -10.2, 95% CI 2-sided [-21.7 to 1.3], Standard Error of Mean 5.841

4. Secondary Outcome: Change in Body Weight (kg) From Baseline to Week 28
Description: Change in body weight (kg) from baseline to Week 28/Study Termination.
Time Frame: Baseline to Week 28
Population: Modified Intent-to-Treat: Subjects who were randomized and received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Experimental: Exenatide QWS Suspension | Active Comparator: Exenatide BID
Number analyzed (Participants) | 229 | 146
kg | -1.49 (0.2842) | -1.89 (0.3640)
Statistical Analysis 1: Comparison: Experimental: Exenatide QWS Suspension vs Active Comparator: Exenatide BID; Test type: Superiority or Other; p = 0.3744, Cochran-Mantel-Haenszel; LS Mean Difference = 0.40, 95% CI 2-sided [-0.48 to 1.28], Standard Error of Mean 0.4497

5. Secondary Outcome: Change in 2-hour Postprandial Glucose Concentrations From Baseline to Week 16
Description: Change in 2-hour postprandial glucose concentrations from baseline to Week 16.
Time Frame: Baseline to Week 16
Population: Meal Test Evaluable Subjects: Subjects who were randomized and received at least one dose of study drug and who participated in the meal test at Visit 3 and Visit 13, had adequate and reliable data for the postprandial data evaluation, and had adequate study medication exposure.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Experimental: Exenatide QWS Suspension | Active Comparator: Exenatide BID
Number analyzed (Participants) | 37 | 31
mg/dL | -87.00 (12.8374) | -113.74 (14.8042)
Statistical Analysis 1: Comparison: Experimental: Exenatide QWS Suspension vs Active Comparator: Exenatide BID; Test type: Superiority or Other; p = 0.0985, Cochran-Mantel-Haenszel; LS Mean Difference = 26.74, 95% CI 2-sided [-5.16 to 58.64], Standard Error of Mean 15.8957

ADVERSE EVENTS:
Time Frame: up to 52 week data reported
Arm/Group | Experimental: Exenatide QWS Suspension | Active Comparator: Exenatide BID
Serious Adverse Events (participants affected / at risk) | 12/229 | 17/146
Other Adverse Events (participants affected / at risk) | 121/229 | 94/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Exenatide QWS Suspension (N=229) | Active Comparator: Exenatide BID (N=146)
Localised Infection (Infections and infestations) | 1 (1) | 0 (0)
Salmonellosis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Septic Shock (Infections and infestations) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diverticular Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Toxic Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hidradentis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Drug Withdrawal Syndrome (General disorders) | 0 (0) | 1 (1)
Lactic Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Umbilical Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Infectious Colitis (Infections and infestations) | 1 (1) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatocellular Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carotid Artery Stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Exenatide QWS Suspension (N=229) | Active Comparator: Exenatide BID (N=146)
Injection Site Nodule (General disorders) | 36 (37) | 6 (6)
Nausea (Gastrointestinal disorders) | 22 (30) | 33 (38)
Headache (Nervous system disorders) | 14 (16) | 9 (10)
Upper Respiratory Tract Infection (Infections and infestations) | 15 (16) | 8 (9)
Diarrhoea (Gastrointestinal disorders) | 14 (23) | 18 (24)
Vomiting (Gastrointestinal disorders) | 9 (11) | 11 (11)
Nasopharyngitis (Infections and infestations) | 11 (13) | 9 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less